CLINICAL TRIAL: NCT06905197
Title: A Phase 1, Open-Label, Multicenter Study to Assess the Safety, Tolerability, Pharmacokinetics, and Anti-tumor Efficacy of DZD6008 in Patients With Advanced Non-small Cell Lung Cancer (NSCLC) With EGFR Mutations (TIAN-SHAN1)
Brief Title: A Multinational Study Assessing an Oral EGFR Inhibitor, DZD6008 in Patients Who Have Advanced NSCLC With EGFR Mutations (TIAN-SHAN1)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Dizal Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: DZ2023C0001
Record Dates: First submitted 2025-03-25; First posted 2025-04-01 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Experimental: Part A Dose Escalation cohorts (20 mg once daily [QD]) (Experimental)
  Interventions: Drug: DZD6008
- Experimental: Part A Dose Escalation cohorts (40 mg QD) (Experimental)
  Interventions: Drug: DZD6008
- Experimental: Part A Dose Escalation cohorts (60 mg QD) (Experimental)
  Interventions: Drug: DZD6008
- Experimental: Part A Dose Escalation cohorts (90 mg QD) (Experimental)
  Interventions: Drug: DZD6008
- Experimental: Part A Dose Escalation cohorts (120 mg QD) (Experimental)
  Interventions: Drug: DZD6008
- Experimental: Part A Dose Escalation cohorts (150 mg QD) (Experimental)
  Interventions: Drug: DZD6008
- Experimental: Part B Dose Expansion cohorts (selected dose 1 QD) (Experimental)
  Interventions: Drug: DZD6008
- Experimental: Part B Dose Expansion cohorts (selected dose 2 QD) (Experimental)
  Interventions: Drug: DZD6008

INTERVENTIONS:
Drug: DZD6008 — Daily dose of DZD6008

SUMMARY:
This study is designed to evaluate safety and anti-tumor activity of DZD6008 in patients with advanced NSCLC with EGFR mutations.

DETAILED DESCRIPTION:
The study includes two parts: Part A (dose escalation) and Part B(dose expansion). In Part A, locally advanced or metastatic NSCLC patients with EGFR sensitizing mutations (Exon19del and/or L858R) following at least 1 prior EGFR TKI regimen will be enrolled. In Part B, locally advanced or metastatic NSCLC patients with EGFR sensitizing mutations following 1 line of the third generation of EGFR TKI treatment will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be able to provide documented informed consent.
2. Aged ≥ 18 years.
3. Histologically or cytologically confirmed diagnosis of NSCLC, locally advanced or metastatic, not suitable for curative therapy.
4. Documentation of EGFR sensitizing mutations (Exon19del and/or L858R) from a local CLIA-certified laboratory (or equivalent).
5. Provide adequate amount of pretreatment tumor samples collected after disease progression on the last EGFR TKI treatment.
6. Failed (progressed or are intolerant) from at least 1 prior EGFR TKI regimen.
7. ECOG 0 or 1 with predicted life expectancy ≥ 12 weeks.
8. Patients with brain metastases must have a stable BM status.
9. Measurable disease per RECIST 1.1.
10. Adequate hematopoietic and other organ system functions.
11. Male Patients with female partners of childbearing potential should use barrier contraceptives and refrain from donating sperm during their participation in this study and for 3 months following the last dose of the study drug.

Exclusion Criteria:

1. Carry any other known EGFR alterations, including but not limited to uncommon EGFR mutations (G719X, S768I, L861Q, exon 20 insertions, etc.)(Part B).
2. NSCLC with mixed small cell lung cancer (SCLC) or NSCLC with histologic SCLC transformation.
3. Prior treatment with any of the following: 1)Immunotherapy or other antibody therapy within 4 weeks prior to the first administration; 2)Any cytotoxic chemotherapy, investigational drugs or other anticancer drugs from a previous treatment regimen or clinical study within 14 days prior to the first administration; 3)Radiotherapy with a limited field of radiation for palliation within 7 days of the first dose, radiation to more than 30% of the bone marrow or with a wide field of radiation within 28 days before screening; 4)Currently receiving or unable to stop drug or herbal supplements known to be potent inhibitors or inducers of cytochrome P450 (CYP)3A4. A washout period of at least 2 weeks for strong inhibitors and 3 weeks for strong inducers is required prior to the first study drug administration; 5)currently receiving or unable to stop drugs known to be CYP3A4 sensitive substrate with a narrow therapeutic index. A washout period of at least 14 days is required prior to the first study drug administration; 6)currently receiving or unable to stop drugs known to be proton pump inhibitors. A washout period of at least 7 days is required prior to the first study drug administration; 7)major surgery within 4 weeks of the first administration of DZD6008 or anticipated during the study period.
4. Any unresolved toxicities from prior anti-cancer therapy greater than CTCAE Grade 1.
5. Spinal cord compression or leptomeningeal metastasis.
6. Patients with any other malignancy within 2 years of the first administration of study drug.
7. Any evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension and active bleeding diatheses as judged by investigator.
8. Patients with active infection, including but not limited to HBV, HCV, HIV and active infection of COVID-19.
9. Resting QTcF > 470 msec; Any clinically significant abnormalities in rhythm, conduction or morphology of resting ECG;Any factors that increase the risk of QTc prolongation.
10. Past medical history of ILD or active ILD.
11. Diseases which would preclude adequate absorption of DZD6008.
12. Received a live vaccine within 2 weeks before the first administration of DZD6008.
13. Women who are pregnant or breastfeeding.
14. Hypersensitivity to active or inactive excipients of DZD6008.
15. Involvement in the planning and conduct of the study.
16. Judgment by the investigator that the patient is unlikely to comply with study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-05-13 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Part A: To assess safety and tolerability | 21 days after the first multiple dose
  Number of participants with Dose-limiting Toxicities (DLTs)
Part A: To assess safety and tolerability | Through the study completion, an average of around 1 year
  Number of participants with Adverse events (AEs)/Serious adverse events (SAEs)
Part B: To assess anti-tumor activity | Through the study completion, an average of around 1 year
  Objective Response Rate (ORR) assessed by Independent Review Committee (IRC) per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1

SECONDARY OUTCOMES:
Part A: To characterize the plasma concentration of DZD6008 following single and multiple oral dose administration | From first dosing to cycle 7 day 1, each cycle is 21 days
  Total concentrations of DZD6008 in plasma
Part A: To assess the anti-tumor activity | Through the study completion, an average of around 1 year
  ORR assessed by investigators per RECIST version 1.1
Part A: To assess the anti-tumor activity | Through the study completion, an average of around 1 year
  Duration of Response (DoR) assessed by investigators per RECIST version 1.1
Part A: To assess the anti-tumor activity | Through the study completion, an average of around 1 year
  Progression Free Survival (PFS) assessed by investigators per RECIST version 1.1
Part B: To assess the anti-tumor activity | Through the study completion, an average of around 1 year
  ORR assessed by investigators per RECIST version 1.1
Part B: To assess the anti-tumor activity | Through the study completion, an average of around 1 year
  DoR assessed by IRC and investigators per RECIST version 1.1
Part B: To assess the anti-tumor activity | PFS assessed by IRC and investigators per RECIST version 1.1
  Through the study completion, an average of around 1 year
Part B: Plasma concentration of DZD6008 | Time Frame: From first dosing to cycle 11 day 1, each cycle is 21 days
  Total concentrations of DZD6008 in plasma
Part B: To assess safety and tolerability | Through the study completion, an average of around 1 year
  Number of participants with AEs/SAEs

CONTACTS AND LOCATIONS:
Locations (5):
- United States (3):
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone Health, New York, New York
  - Herbert Irving Comprehensive Cancer Center, New York, New York
  - Virginia Cancer Specialist (NEXT Oncology-Virginia), Fairfax, Virginia
- Australia (2):
  - Blacktown Hospital, Blacktown, New South Wales
  - Chris O'Brien Lifehouse, Camperdown, New South Wales

IPD SHARING:
Plan to Share IPD: No